CLINICAL TRIAL: NCT04803032
Title: Trident Landmark as a Safe and Easy Method for Facial Nerve Trunk Identification During Superficial Parotidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Collaborators: Fayoum University (Other)
Responsible Party: Principal Investigator, Reda F. Ali, Lecturer of general surgery, Kafrelsheikh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10011616171
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Parotid Tumor; Parotid Neoplasms; Surgery; Head and Neck Disorder
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Superficial parotidectomy using trident landmark technique (Experimental): A modified Blair incision was made along the preauricular skin crease with the same steps of the routine parotid surgery. Dissection was performed using bipolar cautery and blunt instrument; from the tragal cartilage (the anterior surface) until the bony anterior wall of the external auditory canal (EAC); from there, the dissection was done using a blunt instrument. The styloid process's base is the upper point of the trident landmark; it is the superior portion of the trident landmark. Identification of the posterior belly of the digastric muscle till its origin was performed deep to the sternocleidomastoid muscle; it is the lower point of the landmark. The facial nerve is located in the region between these two structures.
  Interventions: Procedure: Superficial parotidectomy

INTERVENTIONS:
Procedure: Superficial parotidectomy — The parotid gland was exposed with its capsule by subplatysmal and SMAS flaps. Dissection was performed from the tragal cartilage until the bony anterior wall of the external auditory canal; from there, the dissection was done using a blunt instrument. The styloid process's base is the upper point of the trident landmark; it is the superior portion of the trident landmark. Identification of the posterior belly of the digastric muscle till its origin was performed deep to the sternocleidomastoid muscle. ); it is the lower point of the landmark. The FNT is located in the region between these two structures. The dissection after identification of the main trunk of the facial nerve was similar to the routine parotidectomy. The surgical defect was closed over a removac suction drain using Vicryl materials; the skin was closed by 6-0 absorbable sutures. A dressing was applied to the surgical site. Then, a gauze was wrapped over the parotid area and secured around the forehead and neck.

SUMMARY:
The parotid has a close relationship with the extra temporal course of the facial nerve. The study aimed to evaluate the accuracy and safety of trident landmark during superficial parotidectomy in the identification of the facial nerve trunk.

DETAILED DESCRIPTION:
A prospective study was conducted between January 2018 and January 2020 at Kafr El-Sheikh university hospital (KUH) and Al Fayoum University Hospital (FUH), Egypt, on 60 patients with benign parotid tumors in the superficial lobe. All patients were subjected to superficial parotidectomy. The outcome was evaluated regarding the clinical success of facial nerve identification by trident landmark and early postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patients with benign tumors of the superficial lobe of the parotid gland

Exclusion Criteria:

* cancers
* unfit patients for surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Number of cases with successful identification of the facial neve by trident landmark | 60 min
  measuring the rate of success of the trident landmark method in identification of the facial nerve during superficial parotidectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Reda F Ali, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided